CLINICAL TRIAL: NCT02527473
Title: Improving Bystander CPR Quality Through Dispatcher-assisted Basic Life Support Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Do Shin, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SNUH-EM-2014-2498
Record Dates: First submitted 2015-08-04; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Out-of-Hospital Cardiac Arrest; Cardiopulmonary Resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Standard Education Group (No Intervention): Control group will receive standard basic life support training for one hour.
- HEROS Group (Experimental): HEROS group will receive the dispatcher-assisted basic life support training that includes standardized video-based CPR education, interactive role-playing with the dispatcher as well as group discussion for one hour.
  Interventions: Other: Dispatcher-Assisted Basic Life Support CPR Education

INTERVENTIONS:
Other: Dispatcher-Assisted Basic Life Support CPR Education — The training program focuses on working in a team with a dispatcher, re-enacting all steps during an emergency call from recognition of cardiac arrest to performing CPR.
  The one hour training session is split into four parts:
  1. Video self-instruction manikin practice (30 min), including a brief introduction to AED.
  2. Practice in pairs (15 min): Role-playing a simulated emergency scenario as the dispatcher and the rescuer
  3. Debriefing (15 min): Questions, answers and reflection
  4. Homework: Information leaflet handed out including at-home tasks such as operating the speakerphone function on the layperson's own phone
  Arms: HEROS Group

SUMMARY:
In an attempt to enhance OHCA survival by increasing bystander CPR rate, this study will assess the effectiveness of the new basic life support with dispatch assistance (DA-BLS) education program through a simulation experiment.

This study aims to determine whether the new DA-BLS program for possible home bystanders is associated with improved CPR quality. We expect home bystanders who were trained with new DA-BLS education program to show better compliance with CPR instructions given by dispatcher via telephone along with improved CPR quality.

DETAILED DESCRIPTION:
Bystander cardiopulmonary resuscitation (CPR) is a crucial component of survival after out-of hospital cardiac arrest (OHCA). Not only the rate of bystander CPR has been associated with higher OHCA survival rate, but the quality of bystander CPR as measured by proportion of correct chest compression and earlier administration has been highly indicative of positive outcomes as well.

However, bystander CPR rates have been reported to be low in many communities due to low access to CPR training. To address this, among many attempts to improve OHCA survival, enhancing bystander CPR rate and quality through dispatcher-assisted CPR (DA-CPR) to the right target group may be an effective and promising approach.

In DA-CPR, the dispatcher on the emergency line provides CPR instruction over the phone. Over-the-telephone CPR instruction was intended to primarily benefit bystanders who have little or no training, but studies have shown that it can also benefit trained bystanders who are in panic in emergency situations to prompt CPR administration. Trained bystanders who received dispatcher assistance during CPR also showed improved CPR quality.

Previous studies reported that 50-81% of OHCA occurs at home. However, the outcome in private homes was very poor compared to outside private home including public places. One possible reason of such lower survival rate may be that the current CPR education programs for home bystanders are inefficient in properly educating home bystanders to provide quality CPR to the patient. In other words, despite the reported benefits of DA-CPR in both trained and untrained bystanders, performing bystander CPR according to phone instruction provided by the dispatcher may not be easy to follow for certain home bystanders such as women and elderly.

According to a recent analysis of 2012 National OHCA Registry, outcomes after OHCA were significantly lower (adjusted odds ratio; 0.36, 95% confidence intervals; 0.18-0.71) in patients who received home bystander CPR with dispatcher assistance than in patients who received either public or who received home bystander CPR without dispatcher assistance. These results suggest that home bystander CPR with dispatcher assistance did not improve the outcomes due to low compliance of CPR instruction and low CPR performance quality by home bystanders. Considering that the in-home OHCA patients are less likely to receive bystander CPR, there needs a new approach to optimize the low compliance rate and CPR quality in possible home bystanders.

ELIGIBILITY:
Inclusion Criteria:

* Female Seoul residents aged between 35-65 years who are primarily a stay-at-home housewife without regular income OR
* Elderly Seoul residents who are older than 65 years old

Exclusion Criteria:

* No prior CPR training

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change of total no flow time at 6 months | Baseline and 6 months

SECONDARY OUTCOMES:
Change of proportion of correct chest compression at 6 months | Baseline and 6 months